CLINICAL TRIAL: NCT02160171
Title: A Multicentre Clinical Evaluation of a Decision Support Algorithm for Neonatal Seizure Detection
Brief Title: ANSeR- The Algorithm for Neonatal Seizure Recognition Study
Acronym: ANSeR
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: University College, London (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Professor Geraldine Boylan, Professor of Neonatal Physiology, University College Cork
Other Study IDs: GB0113UCC
Record Dates: First submitted 2014-02-03; First posted 2014-06-10 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Neonatal Seizures
Keywords: Decision Support Algorithm; Neonatal Seizures; EEG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Term neonates: Term neonates who are undergoing continuous video amplified Electroencephalogram (aEEG)/Electroencephalogram (EEG) monitoring for clinical purposes (e.g. because seizures were suspected, or the neonate is being treated with therapeutic hypothermia). EEGs will be analysed off line by 'Algorithm for Neonatal Seizure Recognition'
  Interventions: Device: Algorithm for Neonatal Seizure Recognition

INTERVENTIONS:
Device: Algorithm for Neonatal Seizure Recognition — Software system for neonatal seizure detection recognition
  Other Names: ANSeR

SUMMARY:
A Multicentre Clinical Evaluation of a Decision Support Algorithm for Neonatal Seizure Detection: ANSeR

DETAILED DESCRIPTION:
This is a multi-centre study. It will be based on routine clinical practice but will also allow for the off-line retrospective application of ANSeR to a well-defined clinical population in order to establish the potential diagnostic utility of the algorithm.

ELIGIBILITY:
Inclusion Criteria:

All term neonates at risk of seizures are eligible for the ANSeR study.

Neonates ≥ 36 weeks gestation will be recruited if:

They have a need for EEG monitoring.

Exclusion Criteria:

Consent of parents not obtained.

Min Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Term neonates who are undergoing continuous video aEEG/EEG monitoring for clinical purposes (e.g. because seizures were suspected, or the neonate is being treated with therapeutic hypothermia)
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To quantify the overall diagnostic accuracy of the Algorithm. | up to 72 hours
  To measure diagnostic accuracy of ANSeR (Algorithm) and clinicians (in routine clinical practice or optimised clinical practice) during the initial up to but not limited to 72 hour period of post-natal EEG monitoring, using an expert panel as the reference standard.

SECONDARY OUTCOMES:
Inappropriate use/non-use of Anti Epileptic Drugs (AEDs) | up to 72 hours
  To quantify the degree and duration of inappropriate use/non-use of AEDs with
  1. the off-line application of the ANSeR algorithm and
  2. routine clinical practice. To compare (a) and (b).
To examine factors that influence diagnostic accuracy in clinical practice. | up to 72 hours
  To examine factors that influence diagnostic accuracy in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Boylan, Professor, Principal Investigator — University College Cork; Janet Rennie, Doctor, Principal Investigator — University College, London
Locations (6):
- Ireland (2):
  - Cork University Maternity Hospital, Wilton, Cork
  - Rotunda Maternity Hospital, Dublin
- University Medical Centre Utrecht, Wilhelmina Children's Hospital, Utrecht, Netherlands
- Karolinska Institutet and University Hospital, Huddinge, Stockholm County, Sweden
- United Kingdom (2):
  - The London and Homerton Hospital, London
  - University College London Hospitals NHS Foundation Trust, London

REFERENCES:
- [Derived] Rennie JM, de Vries LS, Blennow M, Foran A, Shah DK, Livingstone V, van Huffelen AC, Mathieson SR, Pavlidis E, Weeke LC, Toet MC, Finder M, Pinnamaneni RM, Murray DM, Ryan AC, Marnane WP, Boylan GB. Characterisation of neonatal seizures and their treatment using continuous EEG monitoring: a multicentre experience. Arch Dis Child Fetal Neonatal Ed. 2019 Sep;104(5):F493-F501. doi: 10.1136/archdischild-2018-315624. Epub 2018 Nov 24. PMID 30472660